CLINICAL TRIAL: NCT06158061
Title: Assessment of Serum and Tissue Tryptase Levels in Acne Vulgaris Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Magdy Mounir, resident in dermatology department of Sohag Psychiatric hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-11-04MS
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Active Comparator): Patients with acne vulgaris ≥ 18 years old, both male and female patients will be included.
  Interventions: Diagnostic Test: tryptase enzyme level
- control group (Active Comparator): healthy controls without acne vulgaris or other dermatological diseases like psoriasis, vitiligo, DLE
  Interventions: Diagnostic Test: tryptase enzyme level

INTERVENTIONS:
Diagnostic Test: tryptase enzyme level — In serum:
  Three ml blood will be collected from all participants (patients and controls) by aseptic venipuncture into redtop plain glass tubes. Blood samples will be allowed to coagulate during 30-60 minutes. Serum will be obtained by centrifugation at t 1262 g for 10 minutes, aliquoted, and immediately frozen at -20°C until analyzed to determine serum tryptase level. Serum tryptase concentration will be assessed by a commercially available double antibody sandwich enzyme-linked immunosorbent assay (ELISA) kit.
  In tissue:
  Punch skin biopsies of 3mm depth will be taken under local anesthesia from back of Acne vulgaris patients and from matched sites of control subjects. Skin biopsies will be fixed in 10% formalin solution, and submitted to Pathology department in our institute for routine tissue processing by special stain for assessment of tissue tryptase level and number of mast cells tissue biopsy.

SUMMARY:
Acne vulgaris is an inflammatory disorder of pilosebaceous glands. Acne is a highly prevalent inflammatory disease affecting approximately 9.4% of the world's population , and estimated up to 90% among adolescents. By natural course acne starts at 7-12 ages and mostly resolves by the third decade of individuals life .

Mast cells may play important role in maintenance of physiological functions of our body; they also have a role in pathological and inflammatory mechanisms of many diseases. Tryptase is suggested to be important for survival as no tryptase-deficient human subject has yet been reported. Tryptase is mainly synthesized by mast cells but a very low amount may originate in basophil with no interference with total levels of the enzyme. Tryptase is currently considered as a metabolic signaling and effector mediator for acute mast cell degranulation and late phase of allergy and inflammation .

ELIGIBILITY:
Inclusion Criteria:

* Patients with acne vulgaris ≥ 18 years old, both male and female patients will be included.

Exclusion Criteria:

* Patients with the following criteria will be excluded from our study: 1- Pregnancy and breast feeding women. 2- Women on hormonal contraceptions. 3- Patients on topical/systemic treatment for AV during the last 6 months prior to the study. 4- Patients with other dermatological diseases e.g. psoriasis, vitiligo, DLE, etc. 5- Patients suffering from chronic medical illness such as; diabetes mellitus, thyroid disease, and cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-24 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
serum tryptase level | 8 months
  Three ml blood will be collected from all participants (patients and controls) by aseptic venipuncture into redtop plain glass tubes. Blood samples will be allowed to coagulate during 30-60 minutes. Serum will be obtained by centrifugation at t 1262 g for 10 minutes, aliquoted, and immediately frozen at -20°C until analyzed to determine serum tryptase level. Serum tryptase concentration will be assessed by a commercially available double antibody sandwich enzyme-linked immunosorbent assay (ELISA) kit.
tissue tryptase level | 8 months
  Punch skin biopsies of 3mm depth will be taken under local anesthesia from back of Acne vulgaris patients and from matched sites of control subjects. Skin biopsies will be fixed in 10% formalin solution, and submitted to Pathology department in our institute for routine tissue processing by special stain for assessment of tissue tryptase level and number of mast cells tissue biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alanazi MS, Hammad SM, Mohamed AE. Prevalence and psychological impact of Acne vulgaris among female secondary school students in Arar city, Saudi Arabia, in 2018. Electron Physician. 2018 Aug 25;10(8):7224-7229. doi: 10.19082/7224. eCollection 2018 Aug. PMID 30214705
- [Background] Saleh HM, Deif MA, El-Husseiny RM. Assessment of serum interleukin-19 in acne vulgaris patients of different clinical severities. J Cosmet Dermatol. 2021 Sep;20(9):3034-3040. doi: 10.1111/jocd.13977. Epub 2021 Feb 13. PMID 33538078
- [Background] Jusuf NK, Putra IB, Sari L. Differences of Microbiomes Found in Non-Inflammatory and Inflammatory Lesions of Acne Vulgaris. Clin Cosmet Investig Dermatol. 2020 Oct 22;13:773-780. doi: 10.2147/CCID.S272334. eCollection 2020. PMID 33122933
- [Background] Tang L, Yu B, Liao Y, Long S, Yan H, He Q, Li C. Serum Irisin: A Potential Diagnostic Marker for Insulin Resistance in Acne Vulgaris. Indian J Dermatol. 2022 Jul-Aug;67(4):477. doi: 10.4103/ijd.ijd_251_22. PMID 36578741